CLINICAL TRIAL: NCT06789289
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetic Characteristics of TQC2938 in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of TQC2938 in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQC2938-II-01
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQC2938 injection (Experimental): TQC2938 injection is injected subcutaneously every 28 days for a treatment cycle of 52 weeks.
  Interventions: Drug: TQC2938 injection
- TQC2938 injection Placebo (Placebo Comparator): Subcutaneous injection of 0 mg TQC2938 injection solution, with a treatment cycle of every 28 days, for a total of 52 weeks.
  Interventions: Drug: TQC2938 injection Placebo

INTERVENTIONS:
Drug: TQC2938 injection — TQC2938 is a humanized monoclonal antibody that interfering with the signal cascade.
  Arms: TQC2938 injection
Drug: TQC2938 injection Placebo — TQC2938 is a humanized monoclonal antibody that interfering with the signal cascade.
  Arms: TQC2938 injection Placebo

SUMMARY:
The study is a Phase II, multicenter, double-blind, randomized, parallel, placebo-controlled clinical trial designed to evaluate the efficacy, safety, tolerability, and pharmacokinetic characteristics of TQC2938 in patients with moderate to severe Chronic Obstructive Pulmonary Disease (COPD). It is anticipated that 256 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Understand and sign the written informed consent, and comply with the research process schedule during the study period.；
* Be aged 40-80 years inclusive at the time of signing the informed consent form；
* Have a record of COPD diagnosis for at least 12 months prior to screening；
* At screening or after bronchodilator use at the time of the first dose, FEV1 is ≥20% but <80% of the predicted value；
* The FEV1/forced vital capacity (FVC) ratio, measured after the use of bronchodilators at screening or at the time of the first dose, is less than 0.70；
* At screening, the Modified Medical Research Council (mMRC) score is ≥2；
* At screening, the CAT≥10；
* Current smokers or former smokers (who have quit smoking for at least 6 months before Visit 1) with a smoking history of ≥10 pack-years (for example: 20 cigarettes/day for 10 years). At screening, subjects who meet the definition of current smokers will be referred to a smoking cessation clinic；
* A chest X-ray or computed tomography (CT) scan within the 3 months prior to screening or during the screening period (before the first dose of study medication) confirms that there are no other clinically significant pulmonary diseases present apart from COPD.

Exclusion Criteria:

* History of severe allergic reactions or anaphylaxis to biologic agents, or known hypersensitivity to any component of the study drug, or a history of medications or other allergens that the investigator believes would prevent the subject from participating in the study;
* Current or past confirmed diagnosis of asthma;
* History of other clinically significant pulmonary diseases apart from COPD: such as lung cancer, bronchiectasis, sarcoidosis, pulmonary fibrosis, interstitial lung diseases, cystic fibrosis, constrictive bronchiolitis, tuberculosis, or other active pulmonary diseases;
* Evidence of cor pulmonale with right heart failure；
* Diagnosed with α-1-antitrypsin deficiency;
* History of long-term oxygen therapy with >4 L/min;
* When using respiratory assistive oxygen, the subject's oxygen saturation should be ≥89%;
* Undergone lung volume reduction surgery or procedures within the 12 months prior to screening;
* Subjects participating or planning to participate in an intensive COPD rehabilitation program (subjects in the maintenance phase of a rehabilitation program are eligible for this study);
* History of lung transplantation;
* Any infection requiring hospitalization for ≥24 hours and/or treatment with oral, IV, or IM antibiotics within 4 weeks prior to screening or during the screening period;
* Upper or lower respiratory tract infections requiring antibiotic or antiviral medication within 4 weeks prior to screening or during the screening period;
* Moderate to severe COPD exacerbations within 4 weeks prior to screening or during the screening period.
* Received treatment with oral, IV, or intramuscular (IM) corticosteroids (>10 mg/day prednisone or equivalent dose) within 4 weeks prior to starting study medication;
* Received treatment with clinical trial medication, approved biologics (e.g., omalizumab, dupilumab, and/or anti-Interleukin 5 (IL-5) therapies) within 3 months prior to screening or within 5 half-lives of the drug (whichever is longer), or started or changed non-biologic immunomodulatory or immunosuppressive therapies;
* Receiving palliative care due to chronic respiratory disease, cardiovascular disease, endocrine and other systemic diseases, or cancer (e.g., for subjects with a life expectancy <12 months);
* Undergone major surgery within 8 weeks prior to screening or planning to undergo surgery that requires general anesthesia or hospitalization >1 day during the study period;
* Received or planning to receive live attenuated vaccine within 4 weeks prior to screening, during the screening period, or during the study period;
* Known immune deficiency, including but not limited to HIV infection;
* Elevated Aspartate Aminotransferase (AST), Alanine transaminase (ALT), or total bilirubin ≥2.0× the upper limit of normal (ULN) during the screening period;
* At screening, presence of any of the following: positive for hepatitis B surface antigen (HBsAg), positive for both hepatitis C virus antibody (HCV Ab) and hepatitis C virus RNA (HCV-RNA), positive for both specific and non-specific antibodies for syphilis (TP Ab);
* As determined by the investigator, history of illicit drug or drug abuse within the 12 months prior to screening;
* History of malignancy within 5 years prior to screening, except for those with negligible risk of metastasis or death (e.g., with a 5-year overall survival rate >90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin cancer, localized prostate cancer, or ductal carcinoma in situ;
* Presence of any other serious disease or abnormal clinical laboratory test results that, in the opinion of the investigator, would prevent the subject from safely participating in or completing the study；
* Unstable cardiac disease, myocardial infarction, or New York Heart Association Class III or IV heart failure within 12 months prior to screening;
* History or current presence of clinically significant ECG abnormalities, as determined by the investigator, including but not limited to: (1) Atrial fibrillation (AF) with a rapid ventricular rate >120 bpm; (2) Sustained ventricular tachycardia (VT); (3) Bradycardia with a ventricular rate <45 bpm; (4) Mobitz Type II second-degree atrioventricular block and third-degree atrioventricular block (unless a pacemaker or defibrillator has been implanted);
* Corrected QT interval (QTcF) >450 ms for male subjects or >470 ms for female subjects; for subjects with Q wave, R wave, and S wave (QRS) >120 ms, QTcF >480 ms；
* History of ventricular arrhythmias or risk factors for ventricular arrhythmias, such as structural heart disease (e.g., severe left ventricular systolic dysfunction, severe left ventricular hypertrophy with fibrosis), family history of unexplained sudden death or long QT syndrome, or history of sinus bradycardia (ventricular rate <45 beats/min);
* Pregnant or breastfeeding, or planning to become pregnant during the study period or within 12 weeks after the last dose of TQC2938, or female subjects with a positive pregnancy test at screening or randomization.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The annualized incidence rate of moderate to severe acute exacerbations of chronic obstructive pulmonary disease (AECOPD within 24 weeks | Baseline up to week 24
  Within a 24-week period, the number of acute exacerbations of chronic obstructive pulmonary disease (AECOPD) is converted to an annual incidence rate.

SECONDARY OUTCOMES:
Safety and tolerability assessment | Baseline up to week 64
  The incidence and severity of adverse events, adverse reactions, serious adverse events, as well as abnormal clinical laboratory test indicators, vital signs, physical examinations, and 12-lead electrocardiograms.
Within a 52-week period, the number of acute exacerbations of chronic obstructive pulmonary disease (AECOPD) is converted to an annual incidence rate | Baseline up to week 52
  Within a 52-week period, the number of acute exacerbations of chronic obstructive pulmonary disease (AECOPD) is converted to an annual incidence rate.
The change in trough volume of forceful exhalation in the first second (FEV1) (pre-bronchodilator) from baseline after 24 weeks | Baseline up to week 24
  Comparing the difference between the highest FEV1 values at 24 weeks and at baseline for the subjects.
The change in trough FEV1 (pre-bronchodilator) from baseline after 52weeks | Baseline up to week 52
  Comparing the difference between the lowest FEV1 values at 52 weeks and the lowest FEV1 values at baseline for the subjects.
The change in FEV1 from baseline after 52 weeks of bronchodilator use | Baseline up to week 52
  The change in FEV1 from baseline after 52 weeks of bronchodilator use
The annualized incidence rate of severe AECOPD within 52 weeks | Baseline up to week 52
  Within a 52-week period, the number of severe acute exacerbations of chronic obstructive pulmonary disease (AECOPD) is converted to an annual incidence rate.

CONTACTS AND LOCATIONS:
Locations (40):
- China (40):
  - An Hui Chest Hospital, Hefei, Anhui
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peolpe's Hospital Of Chongqing Banan District, Chongqing, Chongqing Municipality
  - Shunde Hospital Of Southern Medical University, Foshan, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Liuzhou municipal liutie central hospital, Liuchow, Guangxi
  - The First People' Hospital Of YuLin, Yulin, Guangxi
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - The second hospital of hebei medical university, Shijiazhuang, Heibei
  - The First Affiliated Hospital of Jiamusi University, Jiamusi, Heilongjiang
  - The First Hospital of Qiqihar, Qiqihar, Heilongjiang
  - Puyang Oilfield General Hospital, Puyang, Henan
  - The First People's Hospital of Xinxiang City, Xinxiang, Henan
  - Yongcheng People's Hospital, Yongcheng, Henan
  - Henan Chest Hospital, Zhengzhou, Henan
  - The second xiangya hospital of central south university, Changsha, Hunan
  - Shaoyang Central Hospital, Shaoyang, Hunan
  - The Affiliated Hospital of Mongolia Medical College, Hohhot, Inner Mongolia
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Jiangxi Provincal People's Hospital, Nanchang, Jiangxi
  - Meihekou Central Hospital, Meihekou, Jilin
  - Siping Central People's Hospital, Siping, Jilin
  - Heze Municipal Hospital, Heze, Shandong
  - Weifang NO.2 People' Hospital, Weifang, Shandong
  - Shanghai JiaoTong University of medicine Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Linfen Central Hospital, Linfen, Shanxi
  - Xi'An International Medicl Center Hospital, Xi’an, Shanxi
  - Affiliated Hospital Of ChengDu University, Chengdu, Sichuan
  - Leshan People's Hospital, Leshan, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The Fourth Central Hospital of Tianjin, Tianjin, Tianjin Municipality
  - The Third People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - Jinhua Municipal Centeral Hospital Medical Group, Jinhua, Zhejiang
  - The First Affiliated Hospitial Of Ningbo University, Ningbo, Zhejiang
  - Taizhou Hospital Of Zhejiang Province, Taizhou, Zhejiang
  - The 2th School of Medicine ,WMU/The 2th affiliated Hospital and Yuying Children's Hospital of WMU, Wenzhou, Zhejiang